CLINICAL TRIAL: NCT04042948
Title: Randomized Controlled Study of Fever Probability, Risk Factors and Preventive Use of Non-steroidal Anti-inflammatory Drugs on Fever After Removal of Drainage Tube After Lumbar Fusion
Brief Title: Clinical Effect of Preventive Use of Tylenol on Fever After Removal of Drainage Tube in Lumbar Fusion Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00006761-M2019299
Record Dates: First submitted 2019-07-13; First posted 2019-08-02 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Lumbar Spinal Stenosis; Lumbar Disc Herniation; Lumbar Radiculopathy
Keywords: lumbar spinal stenosis; lumbar fusion surgery; drainage tube; removal of drainage tube; fever; prevention of fever; preventive use of non-steroidal inflammatory drug
MeSH Terms: conditions — Spinal Stenosis; Intervertebral Disc Displacement; Radiculopathy; Fever | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant
Masking Description: Randomized control parallel
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): preventive use non-steroidal anti-inflammatory drugs to before the removal of drainage tube
  Interventions: Drug: Tylenol
- Control Group (No Intervention): without any intervention when remove the drainage tube

INTERVENTIONS:
Drug: Tylenol — when we decide to remove the drainage tube, we ask the patient to take a pill of tylenol, and another pill in 12h later
  Arms: Experimental Group

SUMMARY:
This study evaluates the influence of Non-steroidal Anti-inflammatory Drugs on preventing fever after the removal of drainage tube in the patients who suffered lumbar fusion surgery, if the outcome turn out positive, the preventive use of non-steroidal anti-inflammatory drugs could decrease the possibility of fever happening when we remove the tube.

ELIGIBILITY:
Inclusion Criteria:

* adult patient
* diagnosis of lumbar spinal stenosis
* perform decompression and fusion surgery and lay a drainage tube
* understand the test and could sign the name

Exclusion Criteria:

* beside the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
the rate of fever after the removal of drainage tube | 24 hours
  we test the temperature of the patient in 24h after the removal of tube, we define fever if the temperature is higher than 37.8 degree

SECONDARY OUTCOMES:
the level of WBC | 24 hours
  we compare the change of the level of WBC of two groups in 24h after the removal of the drainage tube
the level of CRP | 24 hours
  we compare the change of the level of CRP of two groups in 24h after the removal of the drainage tube
the level of ESR | 24 hours
  we compare the change of the level of ESR of two groups in 24h after the removal of the drainage tube
the temperature | 24 hours
  we compare the change of the level of temperature of two groups in 24h after the removal of the drainage tube

CONTACTS AND LOCATIONS:
Overall Officials: Yun Tian, M.D, Principal Investigator — Peking University Third Hospital, Beijing, China
Locations (1):
- Peking University Third Hospital, Beijing, Haidian, China